CLINICAL TRIAL: NCT04846088
Title: A Randomized, Crossover Clinical Study to Characterize Nicotine Pharmacokinetics and Subjective Effects of Nicotine Pouches in Adult Cigarette Smokers
Brief Title: A Study to Characterize Nicotine Pharmacokinetics and Subjective Effects of Nicotine Pouches in Adult Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British American Tobacco (Investments) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BAT2221031
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Product usage order ABICHDGEF (Experimental): Subjects will use each of the 9 products (ABICHDGEF) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order BCADIEHFG (Experimental): Subjects will use each of the 9 products (BCADIEHFG) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order CDBEAFIGH (Experimental): Subjects will use each of the 9 products (CDBEAFIGH) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order DECFBGAHI (Experimental): Subjects will use each of the 9 products (DECFBGAHI) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order EFDGCHBIA (Experimental): Subjects will use each of the 9 products (EFDGCHBIA) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order FGEHDICAB (Experimental): Subjects will use each of the 9 products (FGEHDICAB) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order GHFIEADBC (Experimental): Subjects will use each of the 9 products (GHFIEADBC) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order HIGAFBECD (Experimental): Subjects will use each of the 9 products (HIGAFBECD) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order IAHBGCFDE (Experimental): Subjects will use each of the 9 products (IAHBGCFDE) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order FEGDHCIBA (Experimental): Subjects will use each of the 9 products (FEGDHCIBA) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order GFHEIDACB (Experimental): Subjects will use each of the 9 products (GFHEIDACB) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order HGIFAEBDC (Experimental): Subjects will use each of the 9 products (HGIFAEBDC) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order IHAGBFCED (Experimental): Subjects will use each of the 9 products (IHAGBFCED) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order AIBHCGDFE (Experimental): Subjects will use each of the 9 products (AIBHCGDFE) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order BACIDHEGF (Experimental): Subjects will use each of the 9 products (BACIDHEGF) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order CBDAEIFHG (Experimental): Subjects will use each of the 9 products (CBDAEIFHG) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order DCEBFAGIH (Experimental): Subjects will use each of the 9 products (DCEBFAGIH) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I
- Product usage order EDFCGBHAI (Experimental): Subjects will use each of the 9 products (EDFCGBHAI) during a familiarization period, followed by a 3 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product I

INTERVENTIONS:
Other: Product A — A 4mg nicotine pouch product
Other: Product B — A 7mg nicotine pouch product
Other: Product C — A 7mg nicotine pouch product
Other: Product D — A 7mg nicotine pouch product
Other: Product E — A 7mg nicotine pouch product
Other: Product F — A 7mg nicotine pouch product
Other: Product G — A 7mg nicotine pouch product
Other: Product H — A 7mg nicotine pouch product
Other: Product I — A 7mg nicotine pouch product

SUMMARY:
This study is designed to evaluate plasma nicotine pharmacokinetic (PK) parameters following the use of nicotine pouches in cigarette smokers who have experience with use of smokeless tobacco (SST) [e.g., snus, moist snuff].

DETAILED DESCRIPTION:
Potential subjects will complete screening procedures to assess their eligibility within 45 days prior to enrollment, randomization and confinement.

Following the Screening Visit, eligible subjects will be scheduled for a Day 1 Check-in visit to complete procedures to confirm eligibility. Eligible subjects will be enrolled and begin confinement at the clinical site for 10 days and 9 nights. In addition, on Day 1, subjects will use at least one nicotine pouch (7 mg nicotine) but no more than 3 pouches to familiarize themselves with the investigational product (IP). Subjects will participate in separate Test Sessions for plasma nicotine PK assessment, one for each IP. Each Test Session will last for approximately 3 hours following the start of the IP use, and will include collection of plasma samples for PK assessments prior to, during, and following IP use.

Safety will be monitored throughout the study by the Principal Investigator (PI) (or designee) by assessing adverse events (AEs), vital sign measurements, physical examinations (including an oral examination), and clinical laboratory tests. Mandatory physical and oral examination will be performed as part of end of study or early termination procedures.

The clinical site will attempt to contact all subjects who used at least one IP (including subjects who terminate the study early) using their standard procedures approximately 7 days after the last IP use to determine if any AE has occurred since the last study visit. A return visit may be scheduled for follow-up assessments at the discretion of the PI or an appropriately qualified designee.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete the questionnaire written in English.
2. Generally healthy males or females, 22 to 65 years of age, inclusive, at the time of consent.
3. Body mass index (BMI) within 18.0 to 40.0 kg/m2, inclusive (minimum weight of at least 50.0 kg) at Screening.
4. Healthy, as determined by no clinically significant medical history, physical examination, 12-lead ECG, vital signs, or laboratory (including hematology, clinical chemistry, urinalysis, and serology) findings at Screening, as judged by the PI or designee.
5. Smoke combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length as the primary source of tobacco use.
6. Self-reported use of smokeless tobacco (ST) products (e.g., moist snuff, snus) at least 1 to 2 times in the subject's lifetime prior to screening.
7. Smokes an average of at least 10 cigarettes per day (CPD) and inhale the smoke, for at least 1 year prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the PI or designee.
8. Agrees to smoke the same usual brand (UB) cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand and style currently smoked most frequently by the subject.
9. Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and at Check-in.
10. Positive urine cotinine test (≥ 200 ng/mL) at Screening.
11. Willing to use the IPs during the study period.
12. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to start of each of nine Test Sessions.
13. If female and of non-childbearing potential, must meet one of the following criteria:

    1. Surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion); or
    2. In a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone levels (≥ 40 mIU/mL).
14. If female and of childbearing potential, must agree to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the IP during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

    1. Abstinence from heterosexual intercourse;
    2. Non-hormonal releasing intrauterine device;
    3. Use of a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of the study medication;
    4. For females of < 35 years old only: Hormonal releasing intrauterine device; or
    5. For females of < 35 years old only: Hormonal contraceptives (e.g., oral/transdermal patch/injectable/implant hormonal birth control products).
15. Agrees to an in-clinic confinement of at least 10 days (9 nights).
16. Must be willing to comply with the requirements and restrictions of the study.

Exclusion Criteria:

1. Inability to tolerate at least one 7 mg nicotine pouch for at least 45 minutes during the Product Familiarization Period at Check-in.
2. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI or designee, makes the study subject unsuitable to participate in this clinical study.
3. History, presence of, or clinical laboratory test results indicating diabetes.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI or designee discretion pending approval from the Medical Monitor.
5. History or presence of bleeding or clotting disorders.
6. Presence of gum bleeding and/or abscess, open mouth sores or oral ulcers at Screening or Check-in.
7. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
8. Clinically significant abnormal findings on the vital signs, physical and oral examinations, medical history, or clinical laboratory results, in the opinion of the PI or designee.
9. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at Check-in.
10. History of severe allergic reaction (including anaphylaxis) to any substance, previous status asthmaticus, food allergies/intolerances/restrictions (including mint, wintergreen or spearmint flavoring), or special dietary needs which, in the judgment of the PI or designee, would contraindicate the subject's participation in the study.
11. Requires concomitant treatment with prescription or non-prescription products that contain pseudoephedrine (e.g., nasal/sinus decongestants).
12. Has used medications known to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, desipramine, isoniazid, ketoconazole, miconazole, phenobarbital, rifampin, tranylcypromine, methoxsalen) within (≤) 3 months prior to Check-in and throughout the study.
13. Hemoglobin level is < 12.5 g/dL for females or < 13.0 g/dL for males at Screening.
14. Females who, at Screening or Check-in, have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
15. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Check-in.
16. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at Screening.
17. Self-reported use of any the study IP currently or in the past.
18. Current, regular user (i.e., > 5 times per month) of any tobacco products other than combustible cigarettes or ST within (≤) 6 months prior to screening.
19. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
20. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous attempt within (≤) 30 days prior to the signing the informed consent.
21. Any use of aspirin (≥ 325 mg/day) or anticoagulants within (≤) 30 days prior to the signing the informed consent.
22. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy within (≤) 30 days prior to the signing the informed consent.
23. Whole blood donation within (≤) 8 weeks (≤ 56 days) prior to the signing of informed consent and between Screening and Check-in.
24. Plasma donation within (≤) 7 days prior to the signing of informed consent and between Screening and Check-in.
25. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
26. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing of informed consent in the current study.
27. History of drug or alcohol dependence within (≤)24 months prior to Screening.
28. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol result at Screening or Check-in.
29. Determined by the PI or designee to be inappropriate for this study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
AUCnic 0-180 mins | 0-180 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve (AUCnic) from time zero to 180 minutes after the start of IP use
Cmax | 180 minutes
  Maximum baseline-adjusted plasma concentration of nicotine

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States